CLINICAL TRIAL: NCT04218357
Title: Probenecid as Pharmacotherapy for Alcohol Use Disorder
Brief Title: Probenecid as Medication for Alcohol Use Disorder (PROB)
Acronym: PROB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Assistant Professor, Brown University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1908002524
Record Dates: First submitted 2020-01-01; First posted 2020-01-06 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Probenecid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probenecid (Experimental): 2g probenecid, one pill by mouth once, for one day
  Interventions: Drug: Probenecid or placebo single administration
- matching placebo (Placebo Comparator): Placebo, one pill by mouth once, for one day
  Interventions: Drug: Probenecid or placebo single administration

INTERVENTIONS:
Drug: Probenecid or placebo single administration — study drug administration with alcohol in the laboratory
  Other Names: Probalan

SUMMARY:
The design is a randomized, within-subject, crossover, double-blind, placebo-controlled human alcohol laboratory study with one oral dose of 2g probenecid or placebo administered in two laboratory sessions.

DETAILED DESCRIPTION:
There will be a total of four study visits. Visit 1 is the screening for eligibility (medical and physical examination). On Visits 2 and 3, participants will undergo an alcohol laboratory session with a one week washout period before administering the alternate therapy. The study will conclude at Visit 4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21-70 (inclusive) years; women >7 drinks/week; men >14 drinks/week;
* meet any DSM-5 criteria score for AUD;
* Breath alcohol Content (BrAC)=0.00 at each visit;
* In good health as confirmed by medical history, physical examination and lab tests;
* Willing to adhere to the study procedures;
* Understand informed consent and questionnaires in English at an 8th grade level

Exclusion Criteria:

* Women who are breastfeeding or have a positive urine screen for pregnancy
* CrCl < 60mL/min
* Taking aspirin (salicylates may reduce effect of probenecid)
* Taking penicillin
* Taking methotrexate (may increase concentration)
* Taking other medications that may interact with probenecid
* History of suicide attempts in the last three years
* Current diagnosis of another substance disorder(s) other than nicotine, as assessed by self-reports and urine toxicology screen at baseline
* History of hypersensitivity to sulfa drugs

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina L Haass-Koffler, PHARMD, PHD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tunstall BJ, Lorrai I, McConnell SA, Gazo KL, Zallar LJ, de Guglielmo G, Hoang I, Haass-Koffler CL, Repunte-Canonigo V, Koob GF, Vendruscolo LF, Sanna PP. Probenecid Reduces Alcohol Drinking in Rodents. Is Pannexin1 a Novel Therapeutic Target for Alcohol Use Disorder? Alcohol Alcohol. 2019 Jan 9;54(5):497-502. doi: 10.1093/alcalc/agz054. PMID 31535696
- [Result] Hornbacher R, Gully BJ, Brown ZE, Brown JC, Magill M, Cioe PA, Swift RM, Sanna PP, Haass-Koffler CL. Probenecid as a pharmacotherapy for alcohol use disorder: A randomized placebo-controlled alcohol interaction trial. Alcohol Clin Exp Res (Hoboken). 2024 Dec;48(12):2391-2403. doi: 10.1111/acer.15470. Epub 2024 Oct 29. PMID 39472130

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo, Then Probenecid: Study Drug one pill by mouth once, for one day
  Matching placebo: Placebo
- Probenecid, Then Matching Placebo: 2g probenecid, one pill by mouth once, for one day
  Probenecid
Period: 1st Allocation
Arm/Group | Matching Placebo, Then Probenecid | Probenecid, Then Matching Placebo
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 2nd Allocation (Cross Over)
Arm/Group | Matching Placebo, Then Probenecid | Probenecid, Then Matching Placebo
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Sample: Placebo, then probenecid one pill by mouth once, for one day or Probenecid then placebo one pill by mouth once, for one day
Arm/Group | Overall Sample
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Diagnosis of alcohol use disorder (AUD) by SCID-5 [Count of Participants; unit: Participants]
  no AUD | 9
  Mild AUD | 12
  Moderate AUD | 8
  Severe AUD | 6

OUTCOME MEASURES:

1. Primary Outcome: Stimulant Effects of Alcohol When Co-administered With Drug or Matching Placebo
Description: The stimulant effect of alcohol is assessed using the Biphasic Alcohol Effects Scale (BAES).
  The BAES is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. It consists of 14 items (score) that are rated on a 11-point scale. 7 of the 14 items comprise the stimulation subscale. Individuals are instructed to rate the extent to which alcohol has produced these feelings at the present time from minimum=0 to maximum=10. The subscale of stimulation has a minimum score of 0 (not at all, best outcome) and a maximum score of 70 (high, worse outcome).
  The scale was validated and published: Martin, C. S., Earleywine, M., Musty, R. E., Perrine, M. W. & Swift R. M. (1993). Development and Validation of the Biphasic Alcohol Effects Scale. Alcoholism: Clinical and Experimental Research, 17, 140-146.
Time Frame: Twice at each laboratory session, visits 2 and 3, during the ascending and descending phase of alcohol administration (BrAC).
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Matching Placebo: Placebo, one pill by mouth once, for one day
  Matching placebo: Placebo
- Probenecid: 2g probenecid, one pill by mouth once, for one day
  Probenecid: safety
Arm/Group | Matching Placebo | Probenecid
Number analyzed (Participants) | 35 | 34
scores on scale
  Ascending alcohol BrAC | 28.23 (21.82) | 25.26 (20.66)
  Descending alcohol BrAC | 20.57 (18.95) | 19.56 (20.33)

2. Secondary Outcome: Sedative Effects of Alcohol When Co-administered With Drug or Matching Placebo
Description: The sedative effect of alcohol is assessed using the Biphasic Alcohol Effects Scale (BAES).
  The BAES is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. It consists of 14 items (score) that are rated on a 11-point scale. 7 of the 14 items comprise the sedation subscale. Individuals are instructed to rate the extent to which alcohol has produced these feelings at the present time from minimum=0 to maximum=10. The subscale of stimulation has a minimum score of 0 (not at all, best outcome) and a maximum score of 70 (high, worse outcome).
  The scale was validated and published: Martin, C. S., Earleywine, M., Musty, R. E., Perrine, M. W. & Swift R. M. (1993). Development and Validation of the Biphasic Alcohol Effects Scale. Alcoholism: Clinical and Experimental Research, 17, 140-146.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Matching Placebo | Probenecid
Number analyzed (Participants) | 35 | 34
scores on scale
  Ascending limb of BrAC | 16.02 (14.21) | 16.79 (15.17)
  Descending limb of BrAC | 16.26 (15.27) | 16.50 (15.15)

3. Secondary Outcome: Alcohol Craving
Description: Alcohol craving is assessed using change in the alcohol urge questionnaire (AUQ).
  The Alcohol Urge Questionnaire (AUQ) consists of eight statements about the respondent's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). Drinking refers to various types of alcohol, including beer, wine and liquor. The respondent is asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "strongly disagree" to "strongly agree." Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Minimum score is 7, maximum score is 48. Higher scores reflect greater alcohol craving (worse outcome).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Matching Placebo | Probenecid
Number analyzed (Participants) | 35 | 34
score on scale
  Ascending limb of BrAC | 23.09 (13.23) | 17.24 (10.47)
  Descending limb of BrAC | 19.63 (12.04) | 18.38 (12.29)
Statistical Analysis 1: Comparison: Matching Placebo vs Probenecid; All outcomes were assessed in real-time in the laboratory testing probenecid compared to placebo condition during the alcohol administration procedure; Test type: Superiority; p = 0.05, GEE; Generalized Estimating Equation with standard errors, and an unstructured correlation matrix with medication and time as within-subject factors

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during two laboratory sessions, visits 2 and 3, at which time probenecid and placebo were administered.
Description: We reported any of the following Adverse Events:
  1. All-Cause Mortality in both conditions (none to report)
  2. Serious Adverse Events: in both conditions (none to report)
  3. Other (Not Including Serious) Adverse Events: A table of anticipated and unanticipated events that exceed a frequency threshold (maximum threshold, 5%) within both conditions, grouped by organ system, with number and frequency of such events in each arm/group of the clinical study (none to report)
Arm/Group | Matching Placebo | Probenecid
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT04218357/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04218357/SAP_001.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT04218357/ICF_002.pdf